CLINICAL TRIAL: NCT06258148
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 3 Trial of TG103 Injection Monotherapy Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study of TG103 Injection Monotherapy in Treatment of Type 2 Diabetes Mellitus
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSA1803-010
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- TG103, 7.5 mg (Experimental): TG103 (7.5 mg) will be administered via subcutaneous injection once a week in subjects with type 2 diabetes.
  Interventions: Drug: TG103
- TG103, 7.5 mg placebo (Placebo Comparator): Placebo will be administered via subcutaneous injection once a week in subjects with type 2 diabetes.
  Interventions: Drug: Placebo
- TG103, 15 mg (Experimental): TG103 (15 mg) will be administered via subcutaneous injection once a week in subjects with type 2 diabetes.
  Interventions: Drug: TG103
- TG103, 15 mg placebo (Placebo Comparator): Placebo will be administered via subcutaneous injection once a week in subjects with type 2 diabetes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TG103 — TG103 injection, 7.5mg, 15 mg, SC, once a week
  Arms: TG103, 15 mg; TG103, 7.5 mg
Drug: Placebo — Placebo, SC, once a week
  Arms: TG103, 15 mg placebo; TG103, 7.5 mg placebo

SUMMARY:
This is a randomized, double-blind, placebo-parallel, multicenter phase 3 clinical trial to evaluate the efficacy of TG103 injection 7.5mg and 15mg once a week monotherapy compared with placebo in subjects with type 2 diabetes with poor glycemic control after diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* 1.Subjects have diagnosed with type 2 diabetes according to the Guidelines for prevention and treatment of type 2 diabetes in China (2020 Edition), and have been diagnosed with T2DM for at least 8 weeks before screening;
* 2.Aged 18 to 75 years (inclusive), no gender limitation;
* 3. Body Mass Index (BMI): 18.5≤BMI≤40;
* 4. No hypoglycemic drugs have been used within 8 weeks before screening, and the blood glucose control is poor after diet and exercise therapy alone
* 5.The continuous use of insulin ≤14 days (except gestational diabetes), and/or the types of hypoglycemic drugs used in combination <3 with the continuous use time ≤4 weeks within 1 year (more than 8 weeks) before screening;
* 6.HbA1c must meet the following criteria:

  * Screening: 7.5% ≤ HbA1c ≤ 11.0% (Local laboratory)
  * Baseline: 7.0% ≤ HbA1c ≤ 10.5% (Central laboratory)
* 7.Subjects of childbearing potential must use reliable methods of contraception throughout the study period and at least 3 months after the last dose to avoid pregnancy in female subjects or pregnancy in the male subject's partner;
* 8. Willing and able to accurately use home glucose meter for self-glucose monitoring;
* 9. Be able to understand and follow the trial procedure, voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

* 1. Type 1 diabetes;
* 2. Body weight change more than 5% within 1 month prior to screening;
* 3. Received any of the following medications:

  1. Prior discontinuation of DPP-4 inhibitors or GLP-1 receptor agonists for efficacy, tolerability, and safety reasons;
  2. Systemic glucocorticoid and growth hormone have been used within 8 weeks before screening;
* 4. History of ≥2 episodes of grade 3 hypoglycemia within 6 months prior to screening, or grade 3 hypoglycemia between screening to randomization;
* 5. Acute complications of diabetes, such as diabetic ketoacidosis and hyperglycemic hyperosmolar status, occurred ≥1 time within 6 months prior to screening;
* 6. Severe chronic complications of diabetes (e.g., proliferative diabetic retinopathy, severe diabetic neuropathy, diabetic foot, etc.) within 6 months prior to screening
* 7. History of acute or chronic pancreatitis prior to screening;
* 8. Subjects with clinically significant gastric emptying abnormalities (e.g., gastric outlet obstruction), severe chronic gastrointestinal diseases (e.g., gastroparesis, inflammatory bowel disease, or intestinal obstruction) within 6 months prior to screening, or who have undergone gastrointestinal surgery that affects gastric emptying;
* 9. Any of the following cardiovascular events within 6 months prior to screening: decompensated cardiac insufficiency (NYHA class III or IV); history of unstable angina pectoris, myocardial infarction, coronary artery bypass grafting, or coronary stent implantation; long QT syndrome or prolonged QTcF interval (QTcF: male >450 ms, female >470 ms) on 12-lead ECG; severe arrhythmias that are evaluated by the investigator to be inappropriate for participation in this clinical trial;
* 10. Hemorrhagic stroke or acute ischemic stroke disease occurred within 6 months prior to screening;
* 11. History of psychiatric diseases (such as depression, anxiety, etc.) during screening; or symptomatic gallbladder disease; or history of other diseases that may endanger the safety of the subject and that the investigator deems inappropriate for enrollment;
* 12. Any type of malignant tumor treated or untreated within 5 years prior to screening (except for clinically cured basal cell carcinoma or carcinoma in situ);
* 13. Severe or acute infection within 4 weeks prior to screening, or refractory urinary tract or genital infection within 6 months prior to screening;
* 14. Having a significant blood system disease (e.g., aplastic anemia, myelodysplastic syndrome) or any disease causing hemolysis or red blood cell instability (e.g., malaria) at screening;
* 15. Subjects with thyroid dysfunction that cannot be controlled by a stable drug dose at screening, or with clinically significant abnormalities in thyroid function examination results requiring drug treatment at screening;
* 16. Personal or family history of medullary thyroid cancer (MTC) or type 2 multiple endocrine tumor syndrome at screening;
* 17. Any of the indicators meet the following criteria:
* i. Systolic blood pressure ≥ 160mmHg or diastolic blood pressure ≥ 100mmHg at screening or before randomization;
* ii. Laboratory tests show any of the following abnormalities:

  1. FPG≥13.9 mmol/L;
  2. ALT or AST≥2.5×ULN;
  3. Total bilirubin (TBiL) ≥2.0×ULN;
  4. Triglyceride >5.7 mmol/L;
  5. eGFR<45 mL/(min*1.73 m^2);
  6. Serum amylase and/or lipase ≥3×ULN;
  7. Hemoglobin <100 g/L;
  8. Calcitonin≥50 ng/L(pg/mL);
* iii. Serological examination:

  1. Human immunodeficiency virus antibody or treponema pallidum antibody is positive;
  2. Hepatitis C antibody is positive, and HCV RNA was higher than the lower limit of the detection reference range;
  3. Hepatitis B surface antigen is positive, and the quantitative detection result of HBV DNA was higher than the lower limit of the detection reference range;
* 18. Known allergy to the test drug, Empagliflozin, or related excipients;
* 19. Subjects who have lost more than 400 mL blood due to blood donation or other reasons within 3 months prior to screening;
* 20. Average alcohol intake more than 21 units of alcohol (male)/14 units of alcohol (female) per week within the 3 months prior to screening (1 unit ≈360 mL beer, or 45 mL spirits with 40% alcohol content, or 150 mL wine);
* 21. Subject participated in any drug or medical device clinical study within 3 months prior to screening (except for screening failure);
* 22. Pregnant or lactating female;
* 23. Not suitable for this study in the investigator's opinion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Changes in glycosylated hemoglobin (HbA1c) | Baseline through Week28

SECONDARY OUTCOMES:
Changes in HbA1c | Baseline through Week52
The percentage of HbA1c≤6.5% and the percentage of HbA1c≤7% | Week28 and 52
Change in fasting plasma glucose (FPG) | Baseline through Week 28 and 52
Change in weight | Baseline through Week 28 and 52
Change in 2h-postprandial plasma glucose (2h-PPG) | Baseline through Week 28 and 52
Change in mean 7-point blood glucose curve ， Change in mean postprandial blood glucose increment . | Baseline through Week 28 and 52
Change in blood lipids (triglycerides, total cholesterol, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol) | Baseline through Week 28 and 52
Proportion of subjects receiving remedial therapy | Week 28 and 52
Incidence of adverse events | Week-2 through 52
Blood concentrations of TG103 | Week 0, 4, 8,16, 28,36, 44,52 and 55
The occurrence of TG103 anti-drug antibodies (ADA) and neutralizing antibody (NAb) | Week 0, 4, 8,16, 28,36, 44,52 and 55

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China